CLINICAL TRIAL: NCT03532555
Title: Enteral Zinc to Improve Growth in Infants at Risk for Bronchopulmonary Dysplasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Utah (Other)
Collaborators: Intermountain Research and Medical Foundation (Other)
Responsible Party: Principal Investigator, Bradley Yoder, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102434
Record Dates: First submitted 2018-04-24; First posted 2018-05-22 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-01

CONDITIONS: Infant,Premature; Bronchopulmonary Dysplasia; Growth Failure
Keywords: zinc
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Failure to Thrive | interventions — Zinc Acetate

STUDY DESIGN:
Intervention Model Description: Infants will be stratified by gestational age (23-24 wks, 25-26 wks, 27-29 wks) and then are randomized to receive supplemental oral zinc acetate or no zinc acetate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc plus standard of care (Active Comparator): Infants will receive daily doses of zinc at 2mg/kg from enrollment through 35 6/7 weeks corrected gestational age.
  Interventions: Dietary Supplement: Zinc Acetate
- Standard of care only (Placebo Comparator): Infants will not receive any doses of zinc through 35 6/7 weeks corrected gestational age
  Interventions: Other: No supplemental zinc

INTERVENTIONS:
Dietary Supplement: Zinc Acetate — Zinc Acetate given with elemental zinc dose of 2mg/kg given orally only daily through 35 6/7 weeks corrected gestational age
  Arms: Zinc plus standard of care
Other: No supplemental zinc — Infants will receive standard of care, which is currently no supplemental zinc
  Arms: Standard of care only

SUMMARY:
Multiple factors contribute to growth failure in infants with BPD, including poor nutrient stores, inadequate intake, increased losses, and increased needs. Furthermore, compared to infants without BPD, those with BPD have increased resting metabolic rates and energy expenditure. Growth deficits manifest as lower weight, length, and head circumference, as well as changes in body composition. These deficits precede the development of BPD and persist post-discharge. While similar rates of growth are observed in very low birth weight infants with and without BPD once receiving equal calories, catch up growth does not occur in the BPD group. Thus, early growth deficits remained uncompensated.

After iron, zinc is the most metabolically active trace element in the human body. It has a critical role in growth, through its actions on growth hormone, IGF-1, IGFBP-3, and bone metabolism. Prematurity is a risk factor for zinc deficiency, as 60% of zinc accretion occurs in the third trimester. Impaired intake and absorption or excess excretion can further increase this risk. Finally, periods of rapid growth, as seen in preterm infants, increase the need for zinc.

Biochemically, zinc deficiency is defined by a serum zinc level less than 55mcg/dl. However, while zinc depletion is associated with deficiency, the opposite may not be true. For example, in starving patients, clinical symptoms of zinc deficiency occur during re-feeding, suggesting overall requirements are related to needs, regardless of overall zinc status. This may be the case in preterm infants, who may have a subclinical deficiency despite serum zinc level. Thus, zinc deficiency should be considered in infants with poor growth despite receiving adequate protein and calories.

The objective of this study is to determine whether enteral zinc supplementation leads to improved growth in infants at risk for bronchopulmonary dysplasia (BPD). The investigator's hypothesis is that enteral zinc supplementation in very preterm infants at high risk for BPD will significantly improve growth compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. 23 0/7 to 29 6/7 weeks GA
2. Birth weight 501 to 1000g, inclusive
3. 14 to 28 days of life, inclusive
4. 14 day BPD risk score ≥ 50% for death or moderate-severe BPD, calculated using the algorithm on the Neonatal Research Network website (https://neonatal.rti.org/index.cfm?fuseaction=BPDCalculator.start).-

Exclusion Criteria:

1. Major congenital and/or chromosomal anomalies
2. Inability to reach 80ml/kg/day enteral feeds by 28 days of life

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Growth rate for weight (g/kg/day) from birth to 36+0 weeks corrected gestational age (CGA) | Birth to 36+0 weeks corrected gestational age
  Average daily changes in weight from birth to 36+0 CGA will be calculated and compared between both arms.
Growth rate for weight (g/kg/day) from birth to 40+0 weeks CGA | Birth to 40+0 weeks corrected gestational age
  Average daily changes in weight from birth to 40+0 CGA (or discharge, whichever happens first) will be calculated and compared between both arms.
Growth rate for length (cm/week) from birth to 36+0 weeks CGA | Birth to 36+0 weeks corrected gestational age
  Average weekly changes in length from birth to 36+0 weeks CGA will be calculated and compared between both arms.
Growth rate for length (cm/week) from birth to 40+0 weeks CGA | Birth to 40+0 weeks corrected gestational age
  Average weekly changes in length from birth to 40+0 weeks (or discharge, whichever happens first) CGA will be calculated and compared between both arms.
Growth rate for head circumference (cm/week) from birth to 36+0 weeks CGA | Birth to 36+0 weeks corrected gestational age
  Average weekly changes in head circumference from birth to 36+0 weeks CGA will be calculated and compared between both arms.
Growth rate for head circumference (cm/week) from birth to 40+0 weeks CGA | Birth to 40+0 weeks corrected gestational age
  Average weekly changes in head circumference from birth to 40+0 weeks CGA (or discharge, whichever happens first) will be calculated and compared between both arms.

SECONDARY OUTCOMES:
Measure changes in serum insulin-like growth factor 1 (IGF-1) | Study day 0 to 36 weeks corrected gestational age
  Differences in baseline, 28 days after study intervention initiation, and 36 weeks CGA will be compared between both arms
Measure changes in serum insulin-like growth factor binding protein 3 (IGFBP-3) | Study day 0 to 36 weeks corrected gestational age
  Differences in baseline, 28 days after study intervention initiation, and 36 weeks CGA will be compared between both arms
Measure rates of severe BPD diagnoses at 36+0 weeks CGA | 36+0 weeks corrected gestational age
  Infants will be screened per the NICHD 2001 criteria for severe BPD at 36+0 weeks CGA and these rates will be compared between the two arms.
Measure changes in bone quality per tibial ultrasound | Study day 0 to 36 weeks corrected gestational age
  Differences in baseline, 28 days after study intervention initiation, and 36 weeks CGA will be compared between both arms

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Yoder, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staub E, Evers K, Askie LM. Enteral zinc supplementation for prevention of morbidity and mortality in preterm neonates. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD012797. doi: 10.1002/14651858.CD012797.pub2. PMID 33710626
- [Derived] Vazquez-Gomis R, Bosch-Gimenez V, Juste-Ruiz M, Vazquez-Gomis C, Izquierdo-Fos I, Pastor-Rosado J. Zinc concentration in preterm newborns at term age, a prospective observational study. BMJ Paediatr Open. 2019 Sep 13;3(1):e000527. doi: 10.1136/bmjpo-2019-000527. eCollection 2019. PMID 31646195